CLINICAL TRIAL: NCT07187817
Title: SEquential Treatment of PSoriasis With Biologics
Acronym: STEPS
Status: Recruiting | Type: Observational
Sponsor: Royal United Hospitals Bath NHS Foundation Trust (Other)
Collaborators: University of Bath (Other); University of Leeds (Other)
Responsible Party: Sponsor
Other Study IDs: 001_F_23; 001_F_23 (Other Grant/Funding Number: British Skin Foundation)
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Psoriasis
Keywords: biologic; bdmard; tsdmard; biological agent; 3rd line; 4th line; switch; cycle
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2nd Line Biologic: Participants previously treated with 2 lines of biologic or targeted synthetic treatment for psoriasis.
- 3rd+ Line Biologic: Participants previously treated with 3 or more lines of biologic or targeted synthetic treatment for psoriasis.

SUMMARY:
Psoriasis is a common skin condition that leads to patches of scaled skin which can be inflamed, sore and itchy. It can affect any area of skin on the body, as well as nails, and can be widespread and severe. Over the past 20 years, many new treatments have been developed and approved for severe psoriasis. Most of these newer treatments are given by injection and, as a group, are known as biologics. Many people respond well to biologics and have a meaningful improvement in their condition. There is a smaller proportion of people who do not respond well, or develop side effects, and so must switch drugs to try and improve their condition. In some cases, people need multiple lines of biologic treatment. Currently very little is understood about how well people respond when they are treated with three or more biologics in a row, as very few trials have been done in these cases.

This study aims to use data from people who have already been treated with biologics by their Dermatology teams in the NHS and use the information obtained during their normal clinic appointments to investigate this question. The investigators will assess how well people respond to each line of biologic drug (1st to 10th). They will look at whether people respond as well or less well over time, the more biologics they have. People can be included in the research if they are 18 or over and have been treated with a biologic for psoriasis in participating hospitals in the NHS in England. In this study the investigators are assessing data from events that have previously happened, and so no extra visits are required

DETAILED DESCRIPTION:
STEPS is a retrospective observational cohort study, which will evaluate previously obtained data that had been collected in the process of routine Dermatology appointments. NHS Dermatology centres from around the United Kingdom will be recruited as sites and will submit data on patients with psoriasis treated with biologic drugs (1st to 10th line), from looking through their previous medical notes. All data submitted will be anonymous, as no identifying information will be included in the submissions. An online survey will be developed on the online platform RedCAP to collect and store the data.

Each participant will have information submitted including demographic information like age and sex, as well as information about their psoriasis and treatments. The psoriasis scores (Psoriasis Area and Severity Index and Dermatology Life Quality Index) at baseline of each line of drug, and then at the 3 and 6 month follow up appointments for each line of drug, will be submitted. These measures will be used to determine if there was an improvement in psoriasis with each line of drug, if so what level of improvement, and to compare the response in the different lines of biologic. The hypothesis is that the response at 3 months to each line of biologic does not reduce with increasing lines of biologic after the 2nd line.

As all the information to be submitted has been previously obtained in routine clinics, no additional visits or changes to any medication or monitoring will be required for any participants.

The sample size calculation suggested that a minimum of 610 treatment courses (lines of biologic treatment) are needed to undertake a meaningful analysis, which equates to data on 366 patients. To account for missing data, which is inevitable with observational data, the aim is to recruit 7-8 sites, who will each submit data on 50 patients. The investigators aim for data submission to be completed within 6 months of the start of the study, and that analysis will take a further 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic plaque psoriasis by a Dermatology consultant
* Prior treatment with biologic or targeted synthetic treatment (1 to 10 lines) for psoriasis in the United Kingdom

Exclusion Criteria:

* Diagnosis of other forms of psoriasis for example generalised pustular psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants taken from population who have been treated with biologics and targeted synthetic treatments in Dermatology departments at participating NHS sites.
Sampling Method: Non-Probability Sample
Enrollment: 366 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-02 (Estimated)

PRIMARY OUTCOMES:
PASI75 | 12-16 weeks and 6 months
  75% improvement in Psoriasis Area and Severity Index (PASI)

SECONDARY OUTCOMES:
PASI90 | 12-16 weeks and 6 months
  90% improvement in PASI score
PASI100 | 12-16 weeks and 6 months
  100% improvement to PASI score
PASI<2 | 12-16 weeks and 6 months
  Achievement of a PASI score <2

CONTACTS AND LOCATIONS:
Locations (1):
- Royal United Hospitals Bath NHS Foundation Trust, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD (fully anonymised) would be shared upon reasonable request from other researchers.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT07187817/Prot_SAP_000.pdf